CLINICAL TRIAL: NCT02618980
Title: Management of Acute Upper Gastrointestinal Bleeding in Recent Acute Coronary Syndrome Patients by Early Endoscopy and Non-Endoscopy Treatment: A Randomized Controlled Trial to Evaluate Efficacy and Safety
Brief Title: Early Endoscopy for Acute Upper Gastrointestinal Bleeding in Acute Coronary Syndrome Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment speed due to the incidence of UGI bleeding in ACS patient is lower than expected.
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chen-Shuan Chung, Attending Physician, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-IRB-103062-F
Record Dates: First submitted 2015-11-21; First posted 2015-12-02 (Estimated); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Gastrointestinal Bleeding
Keywords: acute coronary syndrome; gastrointestinal bleeding; endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Acute Coronary Syndrome | interventions — Hemostasis, Endoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early endoscopy (Experimental): endoscopic hemostasis
  Interventions: Other: endoscopic hemostasis
- without early endoscopy (No Intervention): Patients assigned to non-endoscopic treatment group receive high dose infusional PPI therapy. If UGI bleeding subsided after medical treatment alone, diagnostic EGD will be done under stable hemodynamic and 2 weeks after ACS to confirm UGI SRH. If the SRH is not located at UGI tract, the patients will be excluded. Troponin I or T and complete ECG will be checked every 8 hours within 24 hours of interventions. APACHE II score at intervention will be calculated for each patient.

INTERVENTIONS:
Other: endoscopic hemostasis — At endoscopy, stigmata of hemorrhage (SRH) will be treated by dual endoscopic local therapy (combining at least two of the following treatments: epinephrine injection, coaptive thermocoagulation, hemoclip therapy, argon plasma coagulation, bipolar coagulation).
  Arms: early endoscopy

SUMMARY:
The primary aim of this study is to compare efficacy of "early endoscopy" and "non-endoscopic treatment" for management of acute upper gastrointestinal (UGI) bleeding in patients with recent acute coronary syndrome (ACS). This study will also compare rates of surgery, repeated intervention (endoscopy or TAE), rebleeding and complications between two groups.

DETAILED DESCRIPTION:
MATERIALS AND METHODS Study Design and Randomization A multicenter RCT of recent ACS patients presenting with acute UGIB was conducted in three tertiary centers (Far Eastern Memorial Hospital, Hsin-Chu Branch and Taipei Branch of National Taiwan University Hospital) in Taiwan. Patients with recent ACS, including unstable angina (UA), ST-elevation MI (STEMI) and non-ST elevation MI (NSTEMI) who presented symptoms of acute UGIB were evaluated for enrollment. The inclusion criteria were as follows: 1) age over 20-year-old, 2) ACS episodes in the past 2 weeks, 3) symptoms of UGIB including hematemesis, coffee ground emesis or tarry stool passage accompanied with a decrease in hemoglobin (Hb) level greater than 2 g/dl from baseline. Patients with any one of the following criteria were excluded: 1) malignancy or other advanced disease with a life expectancy of < 6 months, 2) pregnant or lactating women, 3) history of allergy or severe side effects from PPIs, contrast, and iodine, 4) platelet count < 80k/uL, or prothrombin time INR >2.0, 5) decompensated (Child-Turcotte-Pugh score B and C) liver cirrhosis, 6) stage 3~5 chronic kidney disease (CKD) (estimated Ccr < 60 ml/min/1.73m2) using Cockcroft-Gault formula, exclusive of end-stage renal disease under renal replacement therapy.17 All the authors had access to the study data and had reviewed and approved the final manuscript.

Eligible patients were randomly assigned to EE or non-EE management. Patients in both groups received bolus intravenous pantoprazole 40mg followed by continuous infusion (8mg/hour).3,18 In the EE group, patients underwent endoscopy within 24 hours after onset of UGIB symptoms. All enrolled patients were monitored in cardiac intensive care unit. At endoscopy, stigmata of hemorrhage (SRH) were treated by endoscopic therapy in combination of any two of the followings: epinephrine submucosal injection, thermocoagulation, hemoclipping, and argon plasma coagulation. Hemostasis was considered initial successful if bleeding had stopped at endoscopy. Antral-biopsy specimens were obtained to a rapid urease test and histopathological examination for Helicobacter pylori (Hp) study. Patients assigned to non-EE group received medical treatment with PPIs alone and underwent esophagogastroduodenoscopy two weeks after enrollment to evaluate the recent SRH. Decision on discontinuation of DAPT was at the discretion of cardiologists depending on cardiac conditions of each enrolled patient.

Study Endpoints The primary endpoint was failure of control hemorrhage. The secondary endpoints included complication rate, length of hospital stay, units of blood transfusion, re-bleeding rate, needs for repeated intervention (endoscopic therapy, transarterial embolization (TAE), or surgery) for uncontrollable recurrent bleeding. Blood troponin-T, creatine kinase-MB, Hb, hematocrit (Hct) and complete electrocardiogram (ECG) were checked every 8 hours within 24 hours after enrollment. APACHE II, Rockall and Blatchford scores at intervention were calculated.19 This study was approved by the Research Ethics Review Committee of study institutes (FEMH IRB-103062-F, Hsin-Chu NTUH 105-001-F, Yun-Lin NTUH 201411020RIND).

Definition of failure to control hemorrhage The time frame for acute bleeding episode was defined as 24 hours after enrollment. Clinical failure of control bleeding was defined as: hematemesis or nasogastric tube drainage of significant fresh blood (≥ 200 mL) ≥ 2hours, or persistent hypovolemic shock after intervention; or 3 g/dl drop in Hb level (or 9% drop of Hct) within 24 hours if no blood transfusion; or a decrease in Hb ≥ 2 g/dL or an increase ≤ 1 g/dL, despite 2 or more units of red blood cells (RBC) component transfusion within 24 hours.

Definition of re-bleeding:

Clinically significant recurrent bleeding was defined by the followings: vomiting of fresh blood, fresh blood in the nasogastric tube aspirate, hematochezia or melena after a normal color stool, and a decrease in Hb ≥ 2 g/dL or an increase less than 1 g/dL, despite 2 or more units of RBC component transfusion.

Definition of major and minor complications Major complications were defined as death and life-threatening arrhythmias within 24 hours after randomization. Minor complications were defined as hypotension (<90/60mmHg), hypertension (>180/100mmHg), tachycardia (>120bpm), bradycardia (<60bpm), tachypnea (>24/min.), oxygen desaturation (SpO2 <90%), and minor arrhythmias.

Sample Size Estimation and Randomization The null hypothesis of this study was the superiority of EE over non-EE in the efficacy on bleeding control. The primary efficacy analysis used an intention-to-treat approach that included all patients meeting the entry criteria who had completed the follow-up. Approximately 80% of UGIB patients will stop bleeding spontaneously,20 and rates of hemostasis that resulted from a first endoscopic procedure exceeded 94% in most large studies.21 However, there was no data demonstrating the outcome of patients under DAPT developing acute UGIB treated medically alone. Therefore, we assumed that about 70% of acute UGIB patients under DAPT would stop bleeding spontaneously without therapeutic endoscopy. As a result, we estimated a sample size of at least totally 78 patients in EE and non-EE groups in order to achieve a statistical power of 80% at a 5% significance level on a two-tailed test, with margin of error of 2% in order to detect a 24% (94% vs. 70%) difference. Sealed envelopes with computer generated randomization number (0 for non-EE, 1 for EE group) were used. After enrollment, gastroenterologists opened the consecutive envelops for randomization.

Statistical Analysis Continuous variables were expressed as mean ± standard deviation and the comparisons between two groups were performed using the Student t-test; categorical variables were summarized as count (%) and the comparisons between groups were made using the Chi-square or the Fisher's exact test when appropriate. Univariate and multivariate logistic regression models were performed for evaluation of the risk factors for outcomes in both groups. A two-tailed p value <0.05 was considered as statistically significant. The statistical analysis was performed using STATA software (version 11.0; Stata Corp, College Station, TX, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent (< 2 weeks) ACS and acute upper GI bleeding accompanied with a decrease in hemoglobin (Hb) level greater than 2 g/dl

Exclusion Criteria (if any one of the following criteria is present):

* Malignancy or other advanced disease with a life expectancy of < 6 months
* Pregnant or lactating women
* History of allergy or severe side effects to PPIs, contrast, and iodine
* Bleeding tendency, and platelet count < 80k/uL, prothrombin time INR >2.0
* Decompensated liver cirrhosis (Child-Pugh classification B~C) and esophagogastric varices history
* Stage 3~5 CKD (estimated Ccr < 60 ml/min/1.73m2) using Cockcroft-Gault formula, exclusive of end-stage renal disease under renal replacement therapy
* Stigmata of hemorrhage confirmed as lower GI tract bleeders
* Without informed consents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Failure of control hemorrhage | 24 hours
  Hematemesis or nasogastric tube drainage of significant fresh blood (≧200 mL) ≧2hours after a specific treatment (therapeutic endoscopy, medical control, transarterial embolization (TAE) or surgery); or Persistent hypovolemic shock; or 3 g/dl drop in Hb level (or 9% drop of Hct) within 24 hours if no transfusion is administered; or A decrease in Hb greater than 2 g/dL or an increase in Hb less than 1 g/dL, despite 2 or more units of blood transfused within 24 hours.

SECONDARY OUTCOMES:
Complication rates | 24 hours
  Major complications are defined as death and life-threatening arrhythmias. Minor complications are defined as hypotension (<90/60mmHg), hypertension (>180/100mmHg), tachycardia (>120bpm), bradycardia (<60bpm), tachypnea (>24/min.), oxygen desaturation (SpO2 <90%), and minor arrhythmias.
length of hospital stay | 14 days
  length of hospital stay
units of blood transfusion | 24 hours
  units of blood transfusion.
re-bleeding rate | 72 hours
  Clinically significant recurrent bleeding was defined by:
  Vomiting of fresh blood, fresh blood in the nasogastric tube aspirate, or hematochezia/melena after normal stool; a decrease in Hb (Hct) greater than 2 g/dL (10%) during any 24-h period, or an increase in Hb (Hct) less than 1 g/dl (3%) for at least 4 units of blood transfused during in 48 hours.
needs for repeated intervention | 72 hours
  endoscopic therapy, angiographic embolization, and surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

REFERENCES:
- [Derived] Chung CS, Chen CC, Chen KC, Fang YJ, Hsu WF, Chen YN, Tseng WC, Lin CK, Lee TH, Wang HP, Wu YW. Randomized controlled trial of early endoscopy for upper gastrointestinal bleeding in acute coronary syndrome patients. Sci Rep. 2022 Apr 6;12(1):5798. doi: 10.1038/s41598-022-09911-5. PMID 35388113